CLINICAL TRIAL: NCT04296760
Title: Rectal Water-contrast Transvaginal Ultrasonography Versus Sonovaginography for the Diagnosis of Posterior Deep Pelvic Endometriosis
Status: Completed | Type: Observational
Sponsor: Fabio Barra (Other)
Responsible Party: Sponsor-Investigator, Fabio Barra, MD, Ospedale Policlinico San Martino
Organization: Ospedale Policlinico San Martino (Other)
Other Study IDs: ENHANCED-ETV-ENDO
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Endometriosis, Rectum; Endometriosis of Vagina; Endometriosis Rectovaginal Septum; Endometriosis Pelvic; Endometriosis of Colon; Endometriosis
Keywords: rectosigmoid endometriosis; posterior pelvic deep endometriosis; vaginal endometriosis; rectovaginal endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with suspicious of deep posterior pelvic endometriosis
  Interventions: Diagnostic Test: Rectal water-contrast transvaginal ultrasonography; Diagnostic Test: Sonovaginography

INTERVENTIONS:
Diagnostic Test: Rectal water-contrast transvaginal ultrasonography — Transvaginal ultrasound scan combined with the introduction of saline solution into the rectum
Diagnostic Test: Sonovaginography — Transvaginal ultrasound scan combined with the introduction of saline solution into the vagina

SUMMARY:
As the surgical treatment of posterior deep endometriosis may be challenging for surgeons and carry significant risks for patients, preoperative assessment of the location, characteristics and presence of nodules of posterior deep endometriosis is important in order to inform the patient about the various treatment possibilities and to allow adequate counseling regarding treatment strategy. The aim of this study is to investigate the accuracy of rectal water-contrast transvaginal ultrasonography (RWC-TVS), and sonovaginography (SVG) in patients with clinical suspicion of posterior deep endometriosis (DIE).

ELIGIBILITY:
Inclusion Criteria:

* clinical presentation suggestive of the presence of posterior deep infiltrating endometriosis

Exclusion Criteria:

* previous diagnosis of posterior deep infiltrating endometriosis by radiologic imaging (i.e. magnetic resonance, computed tomography)
* previous surgical diagnosis of posterior deep infiltrating endometriosis

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patients with suspicion of posterior deep infiltrating endometriosis, referring to our academic department for diagnostic purposes
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Accuracy in diagnosing the presence of the following sites of posterior deep endometriosis: rectovaginal septum, rectosigmoid, uterosacral ligaments, and vagina | At maximum 6 months before undergoing laparoscopic surgical approach

SECONDARY OUTCOMES:
Accuracy in estimating the deep of infiltration in the intestinal muscolari propria of nodules of rectosigmoid endometriosis | At maximum 6 months before undergoing laparoscopic surgical approach
Accuracy in estimating the distance between rectosigmoid endometriosis nodules and the anal verge | At maximum 6 months before undergoing laparoscopic surgical approach
Accuracy in diagnosing the presence of multifocal rectosigmoid endometriosis | At maximum 6 months before undergoing laparoscopic surgical approach
Accuracy in estimating the largest diameter of endometriosis nodules in the following sites of posterior deep endometriosis: rectovaginal septum, rectosigmoid, uterosacral ligaments, and vagina | At maximum 6 months before undergoing laparoscopic surgical approach

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Barra, MD, Principal Investigator — Ospedale Policlinico San Martino
Locations (1):
- Ospedale Policlinico San Martino, Genoa, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leone Roberti Maggiore U, Biscaldi E, Vellone VG, Venturini PL, Ferrero S. Magnetic resonance enema vs rectal water-contrast transvaginal sonography in diagnosis of rectosigmoid endometriosis. Ultrasound Obstet Gynecol. 2017 Apr;49(4):524-532. doi: 10.1002/uog.15934. PMID 27060846
- [Background] Ferrero S, Biscaldi E, Vellone VG, Venturini PL, Leone Roberti Maggiore U. Computed tomographic colonography vs rectal water- contrast transvaginal sonography in diagnosis of rectosigmoid endometriosis: a pilot study. Ultrasound Obstet Gynecol. 2017 Apr;49(4):515-523. doi: 10.1002/uog.15905. PMID 26935873